CLINICAL TRIAL: NCT06296719
Title: Empowering Family Members of Older Adults with Multi-morbidity in Advance Care Planning Conversations: Development and Feasibility Testing of the Chit-Chat Educational Intervention
Brief Title: The Chit-Chat Educational Intervention to Promote Advance Care Planning in the Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ACP Community 2024
Record Dates: First submitted 2024-02-27; First posted 2024-03-06 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-02

CONDITIONS: Old Age; Family Members
Keywords: Family members; Older Adults with multi-morbidity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chit-Chat (Experimental): The Chit-Chat intervention, covering five areas, including (1) Serious illness in older adults, (2) Realities of caring and dying from a carer's perspective, (3) Introduction to the importance of advance care planning for individuals and communities, (4) Effective communication between older adults, family members, and healthcare professionals in ACP conversations (i.e. listening to the wishes and preferences of older adults regarding their needs), and (5) audience participation and clarification including questions, answers and concerns.
  Interventions: Other: Chit-Chat
- Waitlist Control (No Intervention): No intervention

INTERVENTIONS:
Other: Chit-Chat — Participants will receive the 2 sessions of the Chit-Chat intervention on a weekly basis.
  Arms: Chit-Chat

SUMMARY:
The purpose of this study is to estimate the effect size of the Chit-Chat intervention on ACP engagement among family members of older adults with multi-morbidity.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all eligible participants will be asked to provide written informed consent for study entry. At week 0, participants will be randomized in an assessor-blinded randomized controlled trial in a 1:1 ratio to received the Chit-Chat intervention (two 2-hr weekly educational sessions) or wait-list control group.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or above;
* a family member of a relative who aged 60 or above and lives with at least two severe chronic diseases such as cancer, dementia, lung, heart, liver, and renal disease.
* they perceived themselves will take part in taking care of their relatives in the near future;
* able to read and communicate in Cantonese.
* they are self-reported as cognitively intact

Exclusion Criteria:

* their relatives have been referred to palliative care service before the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
ACP engagement | 2 Weeks; 1-month follow-up
  The validated Chinese version of the ACP Engagement Survey - Surrogate Decision Maker consists of 17 items covering 4 dimensions: role cognition, contemplation, self-efficacy, and readiness. The questionnaire used a 5-point Likert scale to gather response. The total score can range between 17 and 85, with higher score indicating higher level of ACP engagement.

SECONDARY OUTCOMES:
Knowledge of ACP | 2 Weeks; 1-month follow-up
  The Knowledge Questionnaire consists of five items which address the purposes of ADs, EOL discussion, and issues related to ACP. The possible range of the total score is 0-5, with higher scores indicating better knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: Doris YP Leung, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Individual participant data are not readily shared because permission to use the data by other researchers has to seek approval from the ethical committee. Request to access IPD should be directed to PI for further consideration and seeking approval from ethical committee.